CLINICAL TRIAL: NCT00338741
Title: Rebif® Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: EMD Serono (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23888
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2010-06-02 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Rebif exposed pregnancies
- 2: Non-Rebif exposed pregnancies

SUMMARY:
The objective for establishing the Rebif® Pregnancy Registry is to collect prospective outcomes data on women in the United States and Canada who have been exposed to Rebif® during their pregnancies. The primary end point will be the rate of spontaneous abortions in exposed pregnancies. This rate will be compared with the rate of spontaneous abortions in patients with Multiple Sclerosis (MS) whose pregnancies were not exposed to any interferon-beta in a manner consistent with the FDA August 2002 Guidance for Industry: Establishing Pregnancy Exposure Registries

DETAILED DESCRIPTION:
This study is a post-approval commitment to follow Rebif®-exposed pregnancies and compare them to non-Rebif® exposed pregnancies to evaluate rate of spontaneous abortion, fetal abnormality or pregnancy related health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Rebif®-Exposed Group

For prospective follow-up, women in the United States and Canada shall be eligible for enrollment in the Rebif® Pregnancy Registry as subjects if:

* They are pregnant.
* They received Rebif® for treatment of Multiple Sclerosis (MS) within one week before or at any time after conception.
* The outcome of pregnancy has not been previously evaluated by any diagnostic method such as ultrasound. However, since ultrasound techniques are often used at early stages to confirm pregnancy, patients who have been evaluated by ultrasound for the purpose of confirming the pregnancy shall be eligible for enrollment in the Registry. The use of ultrasound and any inferences that could be made about the outcome of the patient's pregnancy will be reported on the case report form. Following enrollment in the Registry, diagnostic tests may be performed at any time during the pregnancy.
* They have not used Copaxone® for treatment of MS within the previous three months and have not been exposed to Novantrone®, Imuran®, Cytoxan®, Tysabri® or methotrexate at any time.

Patients who have been exposed to an investigational product or procedure within the previous year may be enrolled at the discretion of the Medical Director. The enrolling physician should contact Serono's authorized agent, a company called Registrat, at 866-997-3243 to request a review of each patient's situation.

Interferon-beta -Not Exposed Comparison Group

Women with MS who live in the United States or Canada will be eligible for the comparison group if:

* They are pregnant.
* The outcome of pregnancy has not been previously evaluated by any diagnostic method such as ultrasound. However, since ultrasound techniques are often used at early stages to confirm pregnancy, patients who have been evaluated by ultrasound for the purpose of confirming the pregnancy shall be eligible for enrollment in the Registry. The use of ultrasound and any inferences that could be made about the outcome of the patient's pregnancy will be reported on the case report form. Following enrollment in the Registry, diagnostic tests may be performed at any time during the pregnancy.
* They have not received any interferon-beta within 90 days of conception.
* They have not used Copaxone® for treatment of MS within the previous three months and have not been exposed to Novantrone®, Imuran®, Cytoxan®, Tysabri® or methotrexate at any time.

Patients who have been exposed to an investigational product or procedure within the previous year may be enrolled at the discretion of the Medical Director. The enrolling physician should contact Serono's authorized agent, a company called Registrat, at 866-997-3243 to request a review of each patient's situation.

Exclusion Criteria:

* Not Applicable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant MS patients
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2002-12; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Mikol, MD, Study Director — EMD Serono
Locations (1):
- Local Medical Information Office, Rockland, Massachusetts, United States

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 physicians in clinical practice in the United States participated in the Registry. Physicians were practicing obstetricians and neurologists who evaluated the subjects as part of their clinical practices.Between 30 Sep 2002 to 15 Feb 2008, 207 subjects were contacted about the Registry. Enrollment was terminated on 07 Dec 2007.
Groups:
- Rebif Exposed Pregnancies: Women with multiple sclerosis (MS) who were exposed to Rebif (interferon-beta [IFN-beta]-1a) during pregnancy or within one week of conception
- Non-Rebif Exposed Pregnancies: Women with MS who had not received any IFN-beta therapy during pregnancy or within 90 days of conception
Period: Overall Study
Arm/Group | Rebif Exposed Pregnancies | Non-Rebif Exposed Pregnancies
Started | 34 (2 subjects signed a consent form but no data were received for either subject) | 2
Completed | 32 | 2
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebif Exposed Pregnancies | Non-Rebif Exposed Pregnancies | Total
Number analyzed (Participants) | 34 | 2 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 33 | 2 | 35
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 2 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 2 | 36

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Abortion
Description: Number of participants having spontaneous abortion
Time Frame: Up to 9 months
Population: Population includes all subjects for whom data is available
Measure: Number; unit: Participants
Arm/Group | Rebif Exposed Pregnancies | Non-Rebif Exposed Pregnancies
Number analyzed (Participants) | 32 | 2
Participants | 2 | 0

2. Secondary Outcome: Fetal Death/Stillbirth
Description: Fetal death/stillbirth
Time Frame: Up to 10 months
Measure: Number; unit: Participants
Arm/Group | Rebif Exposed Pregnancies | Non-Rebif Exposed Pregnancies
Number analyzed (Participants) | 32 | 2
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From study entry until pregnancy outcome. For the purposes of this Registry, the protocol captured as adverse events only unexpected pregnancy events.
Description: These events included spontaneous abortion, stillbirth, elective abortion, anomalies diagnosed at birth, termination or the 28-day follow-up evaluation, labor/delivery complications, pre-eclampsia/eclampsia, premature labor/delivery, and "other" to be specified by the Investigator.
Arm/Group | Rebif Exposed Pregnancies | Non-Rebif Exposed Pregnancies
Serious Adverse Events (participants affected / at risk) | 10/32 | 0/2
Other Adverse Events (participants affected / at risk) | 0/32 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebif Exposed Pregnancies (N=32) | Non-Rebif Exposed Pregnancies (N=2)
Premature labor/premature delivery (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) — Two subjects had premature labor, 1 resulting in a premature delivery and the other in a stillbirth
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Failed induction (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) — 1 for a post-date pregnancy and 1 for an SGA infant.
Failed labour progression (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Uterine fibroids (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Despite a consistent and exhaustive expenditure of resources over 5 years only 36 subjects were enrolled into the Registry, a number which precludes meaningful statistical analysis of the potential risks of Rebif® during pregnancy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other